CLINICAL TRIAL: NCT00303446
Title: Phase II Clinical Trial to Examine the Efficacy and Safety of Dutasteride in Patients With Kennedy's Disease (Spinal and Bulbar Muscular Atrophy)
Brief Title: Dutasteride to Treat Spinal and Bulbar Muscular Atrophy (SBMA)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Kenneth H. Fischbeck, M.D./National Institute of Neurological Disorders and Stroke, National Institutes of Health
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 060113; 06-N-0113 (Other: NINDS IRB protocol number)
Record Dates: First submitted 2006-03-15; First posted 2006-03-16 (Estimated); Results first posted 2010-06-22 (Estimated); Last update posted 2011-01-27 (Estimated); Status verified 2011-01

CONDITIONS: Kennedy's Disease; Spinal and Bulbar Muscular Atrophy
Keywords: Motor Neuron; Androgen Receptor; Polyglutamine; X-Linked; Ligand Dependency; Spinal and Bulbar Muscular Atrophy; SBMA; Kennedy Disease
MeSH Terms: conditions — Bulbo-Spinal Atrophy, X-Linked | interventions — Dutasteride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dutasteride (Active Comparator): Dutasteride 0.5 mg/day
  Interventions: Drug: Dutasteride
- Placebo (Placebo Comparator): Matched placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dutasteride — Dutasteride 0.5 mg/day
  Other Names: Avodart
  Arms: Dutasteride
Drug: Placebo — Matched placebo
  Arms: Placebo

SUMMARY:
This study will determine if the drug dutasteride can improve weakness, mobility, functioning, nerve function, and quality of life in patients with spinal and bulbar muscular atrophy (SBMA). Patients with this inherited disease have an abnormal androgen receptor protein. The male hormones testosterone and dihydrotestosterone (DHT) bind to this abnormal receptor, causing damage to nerve cells that innervate muscle and leading to weakness. Dutasteride decreases DHT production. Lowering DHT levels may decrease the harmful effects of DHT to the nerves and improve strength in people with SBMA.

Males 18 years of age and older with SBMA who have neurological symptoms and can walk 100 feet (with or without assistive devices) may be eligible for this study. Candidates are screened with a blood test and a review of their medical records and genetic studies.

Participants undergo the following procedures:

* Blood and urine tests, history and physical examination, assessment of muscle strength
* Quality-of-life questionnaire
* Tests to assess functional abilities, such walking up steps, keeping the head up while lying down, and other measures
* Nerve conduction study and motor unit number estimation to assess nerve damage. A probe placed on the skin delivers small electrical impulses and wires taped to the skin record the impulses.
* Quantitative muscle testing to measure strength. The subject pushes and pulls levers attached to a gauge. Strength is recorded by a computer.
* Medication. Participants are divided into two groups. One group is given the study drug, dutasteride; the other receives a placebo (sugar pill). All participants take their assigned medication once a day for 24 months.
* Follow-up evaluations. Every 6 months for 2 years, participants return to NIH to repeat the tests described above to determine the effects of the dutasteride. Nerve and quantitative muscle testing is not done at the 6- and 18-month visits.
* In addition to their follow-up appointments here at the NIH every 6 months, participants will also have blood tests and a physical examination performed after 3, 9, 15 and 21 months of treatment by the patient's local physician.

DETAILED DESCRIPTION:
Background:

Spinal and bulbar muscular atrophy (SBMA) or Kennedy's disease is a slowly progressive, X-linked motor neuron disease for which there is currently no treatment. It is caused by a mutation in the androgen receptor that results in a polyglutamine repeat expansion. Recent animal studies have demonstrated that decreasing endogenous androgen levels leads to functional improvement and increased survival. Studies have also shown that high levels of 5 alpha-reductase, the enzyme that converts testosterone to the more potent dihydrotestosterone (DHT), are present in the ventral spinal cord, while low levels of this enzyme are found within skeletal muscle. Thus, by selectively decreasing levels of DHT with dutasteride, a 5 alpha-reductase inhibitor, it is hypothesized that there will be a selective protection of motor neurons, without the adverse effects of reducing the anabolic effects of androgen on muscle.

Objective:

This will be a phase II, double-blind, placebo-controlled trial examining the safety and efficacy of the 5 alpha-reductase inhibitor dutasteride in inhibiting the progression of neurodegeneration in patients with Kennedy's disease. Natural history data will also be obtained from the placebo control arm.

Study Population:

We aim to enroll 50 men with genetically confirmed Kennedy's disease.

Design:

Our objective is to examine the safety and efficacy of dutasteride given at a dose of 0.5 mg a day for 2 years in an outpatient setting. This will be a randomized, double-blind, placebo-controlled trial with 25 subjects in each arm. The subjects will be evaluated neurologically and endocrinologically every 6 months at the NIH Clinical Center. In addition to their clinical visits at the NIH, subjects will also be examined by their primary physician after 3, 9, 15, and 21 months of treatment. The primary objective is to examine the effects of dutasteride on inhibiting or reversing the rate of progression of weakness as measured by quantitative muscle testing. Following informed consent, patients will undergo an initial medical history and physical followed by testing of specific neurological and endocrinological measures over a two-day outpatient visit. Patients will provide blood samples for analysis of hormonal levels and extent of muscle damage every three months. In addition, at the initial, one-year, and two-year follow-up visits patients will have nerve conduction studies as well as quantitative and functional strength evaluation. Each patient will be randomized to the treatment or placebo arm and will be given a 3 month supply of the study drug or a matched placebo at each visit. In between clinic visits, the NIH clinical pharmacy will send an additional 3 month supply to each subject until the subsequent visit.

Outcome Measures:

The primary outcome measure used will be quantitative muscle testing (QMT). Secondary outcome measures include the Adult Myositis Assessment Tool (AMAT), 2-minute walk, a quality of life measure (Medical Outcomes Study 36-item Short Form Version 2, SF-36v2), neurophysiological testing (sensory nerve action potentials, and statistical motor unit number estimation). Changes in hormone levels (testosterone, dihydrotestosterone, androstenedione, estradiol), and creatine kinase levels will also be measured and correlated with changes in strength. Evaluation of disease severity and course as related to CAG repeat length and androgen levels will also be assessed.

Future Directions:

The results of this phase II study will assist us in developing a multi-center, double-blind, placebo-controlled phase III trial. In addition, natural history data will be obtained from the control arm that will be important in future clinical trials of SBMA.

ELIGIBILITY:
Inclusion Criteria:

* Genetically confirmed SBMA
* Neurological symptoms of SBMA
* Ability to ambulate 100 feet with or without the use of assistive devices
* Willingness to participate in all aspects of trial design and follow-up
* Male sex

Exclusion Criteria:

* Age less than 18 years
* Female sex
* A history of hypersensitivity to dutasteride or 5 alpha-reductase inhibitors.
* Exposure to 5 alpha-reductase inhibitors, anti-androgens, testosterone, or steroids in the preceding 6 months
* Patients who are taking potent cytochrome P450 3A4 (CYP3A4) inhibitors for over 4 weeks
* Patients with any pre-existing liver disease
* Alkaline phosphatase, gamma glutamyl transferase, or direct bilirubin greater than 1.5 times the upper limit of normal
* Alanine aminotransferase or aspartate aminotransferase greater than 1.5 times upper limit of normal in subjects with normal creatine kinase levels
* Creatinine greater than 1.5 times the upper limit of normal
* Platelet count, white blood cell count or hemoglobin below the lower limit of normal
* Other clinically significant medical disease that, in the judgment of the investigators, would expose the patient to undue risk of harm or prevent the patient from completing the study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2006-03; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Fischbeck, M.D., Principal Investigator — NINDS, NIH
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Result] Rhodes LE, Freeman BK, Auh S, Kokkinis AD, La Pean A, Chen C, Lehky TJ, Shrader JA, Levy EW, Harris-Love M, Di Prospero NA, Fischbeck KH. Clinical features of spinal and bulbar muscular atrophy. Brain. 2009 Dec;132(Pt 12):3242-51. doi: 10.1093/brain/awp258. PMID 19846582
- [Result] Fernandez-Rhodes LE, Kokkinis AD, White MJ, Watts CA, Auh S, Jeffries NO, Shrader JA, Lehky TJ, Li L, Ryder JE, Levy EW, Solomon BI, Harris-Love MO, La Pean A, Schindler AB, Chen C, Di Prospero NA, Fischbeck KH. Efficacy and safety of dutasteride in patients with spinal and bulbar muscular atrophy: a randomised placebo-controlled trial. Lancet Neurol. 2011 Feb;10(2):140-7. doi: 10.1016/S1474-4422(10)70321-5. Epub 2011 Jan 6. PMID 21216197
- [Derived] Harris-Love MO, Fernandez-Rhodes L, Joe G, Shrader JA, Kokkinis A, La Pean Kirschner A, Auh S, Chen C, Li L, Levy E, Davenport TE, Di Prospero NA, Fischbeck KH. Assessing function and endurance in adults with spinal and bulbar muscular atrophy: validity of the adult myopathy assessment tool. Rehabil Res Pract. 2014;2014:873872. doi: 10.1155/2014/873872. Epub 2014 May 5. PMID 24876969
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/detail/B_2006-N-0113.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 57 subjects were evaluated at the National Institutes of Health (NIH) Clinical Center.
Pre-assignment Details: 7 subjects were excluded on the basis of screening blood test abnormalities. 50 subjects were randomized.
Groups:
- Placebo: Matched placebo, one tablet daily
- Dutasteride: Dutasteride 500 micrograms, one tablet daily.
Period: Overall Study
Arm/Group | Placebo | Dutasteride
Started | 25 | 25
Completed | 23 | 21
Not Completed | 2 | 4
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Death | 0 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Dutasteride | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 21 | 42
  >=65 years | 4 | 4 | 8
Age Continuous [Mean (Standard Deviation); unit: years] | 53.5 (9.2) | 51.9 (10.5) | 53.1 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 25 | 25 | 50
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Muscle Strength Change From Baseline
Description: Quantitative muscle assessment (QMA) was done with a fixed frame dynamometer, a strain gauge tensiometer, and a computer-aided acquisition system. Maximal voluntary isometric muscle contractions were measured twice, the average was calculated, and the results were summed over 22 muscle groups (11 on each side). The total force was scaled for body weight and expressed as percent change from baseline. Measurements were performed at 0, 12, and 24 months. The calculated percent changes at 12 and 24 months are shown.
Time Frame: 0, 12, and 24 months
Population: The participants analyzed were those who were available for analysis at 12 and 24 months.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Dutasteride
Number analyzed (Participants) | 23 | 21
percent change
  Muscle Strength Change From Baseline at 12 Months | -2.2 (9.4) | 3.1 (27.1)
  Muscle Strength Change From Baseline at 24 Months | -4.5 (13.5) | 1.3 (24.2)
Statistical Analysis 1: Comparison: Placebo vs Dutasteride; Test type: Superiority or Other; p = 0.28, Generalized estimating equation model; The analysis includes percent change from baseline at 12 and 24 months

2. Secondary Outcome: Creatine Kinase, Change From Baseline
Description: Serum creatine kinase was determined in venous blood samples analyzed at the Department of Laboratory Medicine of the NIH Clinical Center.
Time Frame: 0, 12, and 24 months
Measure: Mean (Standard Deviation); unit: Units/liter
Arm/Group | Placebo | Dutasteride
Number analyzed (Participants) | 23 | 21
Units/liter
  Creatine kinase change at 12 months | -36 (360) | -32 (375)
  Creatine kinase change at 24 months | -19 (494) | -62 (472)
Statistical Analysis 1: Comparison: Placebo vs Dutasteride; Test type: Superiority or Other; p = 0.86, Generalized estimating equation model; The analysis includes change from baseline at 12 and 24 months

3. Secondary Outcome: Manual Muscle Testing, Change From Baseline.
Description: Manual muscle testing was performed using a modified Medical Research Council (MRC) scale (0=worst, 5=best); the average muscle score was based on 22 muscle groups.
Time Frame: 0, 12, and 24 months
Measure: Mean (Standard Deviation); unit: MRC units on a scale
Arm/Group | Placebo | Dutasteride
Number analyzed (Participants) | 23 | 21
MRC units on a scale
  Manual Muscle Testing, Change at 12 months | 0.04 (0.7) | -0.25 (0.8)
  Manual Muscle Testing, Change at 24 months | 0.02 (0.7) | 0.01 (0.5)
Statistical Analysis 1: Comparison: Placebo vs Dutasteride; Comparison of changes from baseline in manual muscle testing results; Test type: Superiority or Other; p = 0.47, Generalized estimating equation model; The analysis includes change from baseline at 12 and 24 months

4. Secondary Outcome: Adult Myopathy Assessment Tool, Change From Baseline
Description: The Adult Myopathy Assessment Tool rates physical function and muscle endurance, with higher scores indicating better performance; it includes 7 timed functional tasks and 6 endurance tasks (0=worst, 45=best).
Time Frame: 0, 12, and 24 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Dutasteride
Number analyzed (Participants) | 23 | 21
units on a scale
  Adult Myopathy Assessment Tool, Change at 12 mos. | -2.2 (3.7) | -0.7 (2.4)
  Adult Myopathy Assessment Tool, Change at 24 mos. | -2.8 (4.2) | -1.5 (3.9)
Statistical Analysis 1: Comparison: Placebo vs Dutasteride; Test type: Superiority or Other; p = 0.13, Generalized estimating equation model; The analysis includes change from baseline at 12 and 24 months

5. Secondary Outcome: Timed 2-minute Walk, Change From Baseline
Description: The subjects did the 2-minute walk in a 50-foot (15.2-meter) corridor three times, and the average distance was calculated. The subjects were allowed to use an assistive device and rest between the trials.
Time Frame: 0, 12, and 24 months
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Placebo | Dutasteride
Number analyzed (Participants) | 23 | 21
meters
  Timed 2-minute Walk, Change at 12 months | 8.1 (29.8) | -0.8 (28.5)
  Timed 2-minute Walk, Change at 24 months | 2.2 (32.6) | -1.6 (29.6)
Statistical Analysis 1: Comparison: Placebo vs Dutasteride; Test type: Superiority or Other; p = 0.46, Generalized estimating equation model; The analysis includes change from baseline at 12 and 24 months

6. Secondary Outcome: Swallow Score Average, Change From Baseline
Description: Modified barium swallow studies were done at 0, 12, and 24 months. Twenty-five domains were assessed, and six were chosen for final analysis based on the abnormal findings in subjects evaluated at baseline: vallecular pooling and repeated-swallow, each assessed with thin liquids, purees, and solids (rated 1-4, abnormal to normal).
Time Frame: 0, 12, and 24 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Dutasteride
Number analyzed (Participants) | 23 | 21
units on a scale
  Swallow Score Average, Change at 12 months | -0.25 (0.4) | 0.06 (0.6)
  Swallow Score Average, Change at 24 months | -0.53 (0.5) | -0.14 (0.5)
Statistical Analysis 1: Comparison: Placebo vs Dutasteride; Test type: Superiority or Other; p = 0.11, Generalized estimating equation model; The analysis includes change from baseline at 12 and 24 months

7. Secondary Outcome: Bulbar Rating Scale, Change From Baseline
Description: The Bulbar Rating Scale includes eight domains each rated on a 1-4 scale, abnormal to normal. The original 8-32 point scale was transformed to a 0-100% scale to represent the responses as percentages.
Time Frame: 0, 12, and 24 months
Measure: Mean (Standard Deviation); unit: percentage of maximum score
Arm/Group | Placebo | Dutasteride
Number analyzed (Participants) | 23 | 21
percentage of maximum score
  Bulbar Rating Scale, Change at 12 months | 5.7 (6.7) | 2.6 (6.8)
  Bulbar Rating Scale, Change at 24 months | 6.4 (5.8) | 3.9 (4.6)
Statistical Analysis 1: Comparison: Placebo vs Dutasteride; Test type: Superiority or Other; p = 0.08, Generalized estimating equation model; The analysis includes change from baseline at 12 and 24 months

8. Secondary Outcome: Sensory Nerve Action Potential Average, Change From Baseline
Description: Nerve conduction studies were done on four sensory nerves (median, ulnar, radial, sural), and the amplitudes of the evoked responses were averaged. Loss of amplitude indicates impairment of conduction.
Time Frame: 0, 12, and 24 months
Measure: Mean (Standard Deviation); unit: microVolts
Arm/Group | Placebo | Dutasteride
Number analyzed (Participants) | 23 | 21
microVolts
  Sensory Nerve Action Potential, Change at 12 mos. | 0 (1) | 0 (1)
  Sensory Nerve Action Potential, Change at 24 mos. | 0 (1) | 0 (1)
Statistical Analysis 1: Comparison: Placebo vs Dutasteride; Test type: Superiority or Other; p = 0.73, Generalized estimating equation model; The analysis includes change from baseline at 12 and 24 months

9. Secondary Outcome: Median Compound Muscle Action Potential, Change From Baseline
Description: Nerve conduction studies were done on the median motor nerve, and the compound muscle action potential amplitude was determined. Loss of amplitude indicates impairment of conduction.
Time Frame: 0, 12, and 24 months
Measure: Mean (Standard Deviation); unit: mVolts
Arm/Group | Placebo | Dutasteride
Number analyzed (Participants) | 23 | 21
mVolts
  Median Motor Action Potential, Change at 12 months | 0.04 (2.15) | 0.52 (2.63)
  Median Motor Action Potential, Change at 24 months | -0.24 (1.84) | 0.24 (1.89)
Statistical Analysis 1: Comparison: Placebo vs Dutasteride; Test type: Superiority or Other; p = 0.37, Generalized estimating equation model; The analysis includes change from baseline at 12 and 24 months

10. Secondary Outcome: Peroneal Compound Muscle Action Potential, Change From Baseline
Description: Nerve conduction studies were done on the peroneal nerve, and the compound muscle action potential amplitude was determined. Loss of amplitude indicates impairment of conduction.
Time Frame: 0, 12, and 24 months
Measure: Mean (Standard Deviation); unit: mVolts
Arm/Group | Placebo | Dutasteride
Number analyzed (Participants) | 23 | 21
mVolts
  Peroneal Motor Action Potential, Change at 12 mos. | 0.16 (1.07) | 0.02 (0.84)
  Peroneal Motor Action Potential, Change at 24 mos. | 0.15 (1.37) | 0.04 (0.81)
Statistical Analysis 1: Comparison: Placebo vs Dutasteride; Test type: Superiority or Other; p = 0.65, Generalized estimating equation model; The analysis includes change from baseline at 12 and 24 months

11. Secondary Outcome: Motor Unit Nerve Estimation, Change From Baseline
Description: Motor unit number estimation (MUNE) was done with a statistical MUNE program, on the abductor pollicis brevis. All subjects were evaluated on the right side unless severe atrophy produced very low compound muscle action potentials; in this case, the left side was investigated or the abductor digiti minimi was substituted. A decrease in MUNE indicates a loss of motor units.
Time Frame: 0, 12, and 24 months
Measure: Mean (Standard Deviation); unit: motor unit number
Arm/Group | Placebo | Dutasteride
Number analyzed (Participants) | 23 | 21
motor unit number
  Motor Unit Nerve Estimation, Change at 12 months | -4.2 (18.9) | -4.2 (18.7)
  Motor Unit Nerve Estimation, Change at 24 months | -2.2 (23.3) | -2.6 (17.5)
Statistical Analysis 1: Comparison: Placebo vs Dutasteride; Test type: Superiority or Other; p = 0.99, Generalized estimating equation model; The analysis includes change from baseline at 12 and 24 months

12. Secondary Outcome: Activities of Daily Living, Change From Baseline
Description: Subjects rated their daily activity with a modified 9-question Activities of Daily Living (ADL) questionnaire (0-4, fully impaired to normal).
Time Frame: 0, 12, and 24 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Dutasteride
Number analyzed (Participants) | 23 | 21
units on a scale
  Activities of Daily Living, Change at 12 months | 0.4 (2.3) | 0.4 (2.8)
  Activities of Daily Living, Change at 24 months | 1.2 (3.3) | 1.1 (4.2)
Statistical Analysis 1: Comparison: Placebo vs Dutasteride; Test type: Superiority or Other; p = 1.0, Generalized estimating equation model; The analysis includes change from baseline at 12 and 24 months

13. Secondary Outcome: Medical Outcomes Study 36-item Short Form Version 2 (SF-36v2) Physical Component Summary, Change From Baseline
Description: Subjects completed the Medical Outcomes Study Short Form Version 2 (SF-36v2), in which they rated their physical quality of life over the preceding 4 weeks. Raw SF-36v2 scores were converted to norm-based scales and component summaries using the scoring code provided by QualityMetric (mean=50, standard deviation (SD)=10).
Time Frame: 0, 12, and 24 months
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Dutasteride
Number analyzed (Participants) | 23 | 21
percent change
  SF-36v2 Physical Component Sum., Change at 12 mos. | -0.9 (6.5) | 2.5 (5.9)
  SF-36v2 Physical Component Sum., Change at 24 mos. | -3.6 (8.4) | 2.1 (6.1)
Statistical Analysis 1: Comparison: Placebo vs Dutasteride; Test type: Superiority or Other; p = 0.014, Generalized estimating equation model; The analysis includes change from baseline at 12 and 24 months

14. Secondary Outcome: Medical Outcomes Study 36-item Short Form Version 2 (SF-36v2) Mental Component Summary, Percent Change From Baseline
Description: Subjects completed the Medical Outcomes Study Short Form Version 2 (SF-36v2), in which they rated their mental quality of life over the preceding 4 weeks. Raw SF-36v2 scores were converted to norm-based scales and component summaries using the scoring code provided by QualityMetric (mean=50, standard deviation (SD)=10), and percent change in the norm-based scale was calculated.
Time Frame: 0, 12, and 24 months
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Dutasteride
Number analyzed (Participants) | 23 | 21
percent change
  SF-36v2 Mental Component Sum., Change at 12 mos. | 0.6 (11.1) | 0.1 (7.9)
  SF-36v2 Mental Component Sum., Change at 24 mos. | 3.3 (9.3) | -3.2 (10.2)
Statistical Analysis 1: Comparison: Placebo vs Dutasteride; Test type: Superiority or Other; p = 0.033, t-test, 2 sided — Generalized estimating equation model showed a significant interaction between time and treatment; therefore a two sample t-test was used at each time point. P-value is given for comparison at 24 months

15. Secondary Outcome: International Index for Erectile Function (IIEF), Change From Baseline
Description: Sexual function was rated using the International Index of Erectile Function (IIEF). The total IIEF score (5-75, worst-best) was reported as the percent maximum (0-100%).
Time Frame: 0, 12, and 24 months
Measure: Mean (Standard Deviation); unit: percent of maximum score
Arm/Group | Placebo | Dutasteride
Number analyzed (Participants) | 23 | 21
percent of maximum score
  IIEF, Change at 12 months | -2.4 (10.2) | -2.1 (11.6)
  IIEF, Change at 24 months | -0.3 (16.4) | -3.5 (6.9)
Statistical Analysis 1: Comparison: Placebo vs Dutasteride; Test type: Superiority or Other; p = 0.61, Generalized estimating equation model; The analysis includes change from baseline at 12 and 24 months

ADVERSE EVENTS:
Time Frame: 24 months
Description: Subjects reported the severity and type of adverse events at each visit.
Arm/Group | Placebo | Dutasteride
Serious Adverse Events (participants affected / at risk) | 2/25 | 5/25
Other Adverse Events (participants affected / at risk) | 23/25 | 23/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=25) | Dutasteride (N=25)
fall requiring hospitalization (Musculoskeletal and connective tissue disorders) | 2 (4) | 2 (2)
cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) — Death from a probable cardiac event.
gastroenteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) — Dehydration requiring hospitalization.
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Subject developed serious respiratory difficulties and was removed from the study.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=25) | Dutasteride (N=25)
cardiac events (Cardiac disorders) | 3 (3) | 1 (1)
constitutional symptoms (General disorders) | 3 (4) | 6 (14)
dermatologic (Skin and subcutaneous tissue disorders) | 3 (3) | 4 (6)
endocrine (Endocrine disorders) | 0 (0) | 2 (2)
ear-nose-throat (General disorders) | 11 (16) | 10 (20)
gastrointestinal (Gastrointestinal disorders) | 5 (8) | 7 (26)
hematologic (General disorders) | 3 (3) | 2 (2)
hepatic (Hepatobiliary disorders) | 0 (0) | 2 (3)
infectious (Infections and infestations) | 12 (312) | 14 (26)
musculoskeletal (General disorders) | 18 (109) | 11 (73)
neurologic (Nervous system disorders) | 15 (34) | 15 (39)
genitourinary (General disorders) | 1 (2) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No